CLINICAL TRIAL: NCT01259414
Title: Comparison of Two Solvents Used With Chemotherapy Agent for Transarterial Chemoembolization of Hepatocellular Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Shi Ming, Prof., Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HCC2011A
Record Dates: First submitted 2010-12-13; First posted 2010-12-14 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: Carcinoma,Hepatocellular; Liver Neoplasms; Survival analysis; treatment outcome; administration drugs; Chemoembolization,; TACE; polyvinyl alcohol; water-soluble contrast mesium; iopamidol; lipiodol; distilled water
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Solvents

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group1 (Experimental): Chemoembolization with solvent with specific gravity less than lipiodol
  Interventions: Other: Solvent with specific gravity less than lipiodol
- group2 (Experimental): Chemoembolization with Solvent with specific gravity equivalent to lipiodol
  Interventions: Other: Solvent with specific gravity equivalent to lipiodol

INTERVENTIONS:
Other: Solvent with specific gravity less than lipiodol — TACE with chemotherapy drugs (EADM 50mg, lobaplatin 50mg, and MMC 6mg)dissolved in distilled water and emulsified lipiodol followed embolization with polyvinyl alcohol particles (PVA)
  Arms: group1
Other: Solvent with specific gravity equivalent to lipiodol — TACE with chemotherapy drugs (EADM 50mg, lobaplatin 50mg, and MMC 6mg)dissolved in water-soluble contrast medium and distilled water,then emulsified with lipiodol followed embolization with polyvinyl alcohol particles (PVA)
  Arms: group2

SUMMARY:
TACE is considered the standard treatment for unresectable HCC and is widely used as a palliative treatment. However there is no consensus of the protocol of TACE.One of the variation is does the stability of the suspension by emulsified the lipiodol and the contrast medium used to dissolve the anticancer agents really effect the survival.Thus the investigators conduct this prospective,randomized controlled study to find out if the different method of preparing chemotheraputic drugs can cause a different survival benefit.

DETAILED DESCRIPTION:
Transcatheter arterial chemoembolization is currently the mainstays of palliative treatments worldwide for patients with unresectable HCC. However there is no standard protocol exists for TACE currently. One of the controversy is does the way of emulsified the anticancer agents and lipiodol to get a high stability suspension really effect the survival rates.

Anticancer drugs play important role in survival benefit. Many studies have innovated different methods to get a high stability suspension of lipiodol and anticancer drugs ,because they think lipiodol can selectively retained in HCC and used as a drug-carrying which allow a slow release of the anticancer drug from lipiodol microdroplets. Thus ,A stability suspension might get a maximize tumor drug uptake,which can caused a more tumor necrosis, and minimize systemic drug levels ,which get a less toxicity, hence survival benefit. While the other researcher think a stability emulsion can't get a positive effect ,such as pharmacokinetic and systematic toxicity of the anticancer drugs, tumor response, biologic response and so on.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients > 18 years and <=70 years of age with a diagnosis of HCC
* BCLC B stage disease
* Not amendable to surgical resection ,local ablative therapy and any other cured treatment.
* Patients must have at least one tumor lesion that can be accurately measured according to EASL criteria. The lesion has not been previously treated with TACE, surgery, radiation therapy, radiofrequency ablation, percutaneous ethanol or acetic acid injection, or cryoablation.
* No Cirrhosis or cirrhotic status of Child-Pugh class A only
* Not pregnant or breast-feeding patients
* No significant renal impairment (creatinine clearance < 30 mL/minute) or patients on dialysis
* The following laboratory parameters:

  * Platelet count ≥ 60,000/µL
  * Hemoglobin ≥ 8.5 g/dL
  * Total bilirubin ≤ 1.5 mg/dL Serum albumin ≥ 35 g/L
  * ASL and AST ≤ 5 x upper limit of normal
  * Serum creatinine ≤ 1.5 x upper limit of normal
  * INR ≤ 1.5 or PT/APTT within normal limits
  * Absolute neutrophil count (ANC) >1,500/mm3
* Ability to understand the protocol and to agree to and sign a written informed consent document

Exclusion Criteria:

* Known history of HIV
* History of organ allograft
* Known or suspected allergy to the investigational agents or any agent given in association with this trial.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Evidence of bleeding diathesis.
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first dose of study drug
* Serious non-healing wound, ulcer, or bone fracture
* Known central nervous system tumors including metastatic brain disease
* severe Arterioportal Shunts or Arteria vein Shunts

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 812 (Estimated)
Dates: Start 2011-01; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
overall survival | 3 year

SECONDARY OUTCOMES:
Time to progression | 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Ming Shi, Principal Investigator — Cancer Center, Sun Yat-set University
Locations (1):
- Cancer Center Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Shin SW. The current practice of transarterial chemoembolization for the treatment of hepatocellular carcinoma. Korean J Radiol. 2009 Sep-Oct;10(5):425-34. doi: 10.3348/kjr.2009.10.5.425. Epub 2009 Aug 25. PMID 19721826
- [Result] Lo CM, Ngan H, Tso WK, Liu CL, Lam CM, Poon RT, Fan ST, Wong J. Randomized controlled trial of transarterial lipiodol chemoembolization for unresectable hepatocellular carcinoma. Hepatology. 2002 May;35(5):1164-71. doi: 10.1053/jhep.2002.33156. PMID 11981766
- [Result] Llovet JM, Real MI, Montana X, Planas R, Coll S, Aponte J, Ayuso C, Sala M, Muchart J, Sola R, Rodes J, Bruix J; Barcelona Liver Cancer Group. Arterial embolisation or chemoembolisation versus symptomatic treatment in patients with unresectable hepatocellular carcinoma: a randomised controlled trial. Lancet. 2002 May 18;359(9319):1734-9. doi: 10.1016/S0140-6736(02)08649-X. PMID 12049862
- [Result] Raoul JL, Heresbach D, Bretagne JF, Ferrer DB, Duvauferrier R, Bourguet P, Messner M, Gosselin M. Chemoembolization of hepatocellular carcinomas. A study of the biodistribution and pharmacokinetics of doxorubicin. Cancer. 1992 Aug 1;70(3):585-90. doi: 10.1002/1097-0142(19920801)70:33.0.co;2-#. PMID 1320447
- [Result] Bruix J, Sherman M; Practice Guidelines Committee, American Association for the Study of Liver Diseases. Management of hepatocellular carcinoma. Hepatology. 2005 Nov;42(5):1208-36. doi: 10.1002/hep.20933. No abstract available. PMID 16250051
- [Result] Takaki Y, Kaminou T, Shabana M, Ihaya T, Otsubo K, Ogawa T. Suitable blending method of lipiodol-cisplatin in transcatheter arterial embolization for hepatocellular carcinoma: evaluation of sustained release and accumulation nature. Hepatogastroenterology. 2008 Jan-Feb;55(81):202-6. PMID 18507107
- [Result] de Baere T, Zhang X, Aubert B, Harry G, Lagrange C, Ropers J, Dufaux J, Lumbroso J, Rougier P, Ducreux M, Roche A. Quantification of tumor uptake of iodized oils and emulsions of iodized oils: experimental study. Radiology. 1996 Dec;201(3):731-5. doi: 10.1148/radiology.201.3.8939223.
- [Result] Takayasu K, Shima Y, Muramatsu Y, Moriyama N, Yamada T, Makuuchi M, Hasegawa H, Hirohashi S. Hepatocellular carcinoma: treatment with intraarterial iodized oil with and without chemotherapeutic agents. Radiology. 1987 May;163(2):345-51. doi: 10.1148/radiology.163.2.3031724.
- [Result] Tzeng WS, Wu RH, Chang SC, Chou CK, Lin CY, Chen JJ, Yang SC, Lin CH. Ionic versus nonionic contrast media solvents used with an epirubicin-based agent for transarterial chemoembolization of hepatocellular carcinoma. J Vasc Interv Radiol. 2008 Mar;19(3):342-50. doi: 10.1016/j.jvir.2007.10.021. PMID 18295692